CLINICAL TRIAL: NCT01580423
Title: The Role of Substance P on Perception of Breathlessness
Brief Title: The Role of Substance P on Perception of Breathlessness During Resistive Load Breathing
Acronym: SP-RLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CPHS23276
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aprepitant (Experimental)
  Interventions: Drug: aprepitant
- inert powder (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aprepitant — 125 mg capsule
  Arms: aprepitant
Drug: placebo — capsule identical to aprepitant
  Arms: inert powder

SUMMARY:
Substance P is released from sensory nerves and transmits pain information into the central nervous system. As pain and dyspnea share many characteristics, including similar neurological pathways, it is possible that substance P may contribute to the sensation of dyspnea. The hypothesis of the study is that patients with chronic obstructive pulmonary disease (COPD) will provide lower ratings of breathlessness during resistive load breathing with oral aprepitant, a medication that blocks the activity of substance P, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* diagnosis of COPD
* former smoker > 10 pack-years
* clinical diagnosis of chronic bronchitis
* post-bronchodilator forced expiratory volume in one second (FEV1) 30 - 80% predicted
* FEV1/forced vital capacity ratio less than or equal to 70%

Exclusion Criteria:

* current smoker
* pregnant women
* concomitant disease that might interfere with study procedures
* peripheral vascular disease or cold hypersensitivity
* drugs that might interfere with aprepitant

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Mahler, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: April to October 2012; Location: medical clinic
Pre-assignment Details: 17 subjects recruited; 1 patient who signed the consent form did not meet inclusion/exclusion criteria, and no testing was performed.
Groups:
- First Aprepitant, Then Inert Powder: Capsule of aprepitant 125 mg in first intervention period and capsule of inert powder in second intervention period.
- First Inert Powder, Then Aprepitant: Capsule of inert powder in first intervention period and capsule of aprepitant 125 mg in second intervention period.
Period: First Intervention
Arm/Group | First Aprepitant, Then Inert Powder | First Inert Powder, Then Aprepitant
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | First Aprepitant, Then Inert Powder | First Inert Powder, Then Aprepitant
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive aprepitant first and inert powder first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 70.2 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Intensity of Breathlessness
Description: Time-weighted averages of intensity of breathlessness.
  Subject rating of intensity of breathlessness was obtained at 1 minute intervals during RLB on a 100 mm Visual Analog Scale anchored at the bottom by "No Intensity" and at the top by "Greatest Intensity".
Time Frame: At 1 minute intervals during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Aprepitant: Capsule containing 125 mg of aprepitant
- Inert Powder: Capsule containing inert powder
Arm/Group | Aprepitant | Inert Powder
Number analyzed (Participants) | 16 | 16
units on a scale | 80.8 (13.5) | 77.9 (14.5)

2. Secondary Outcome: Intensity of Pain
Description: Time-weighted averages for intensity of pain.
  Subject rating of intensity of pain on a 100 mm Visual Analog Scale anchored at the bottom by "No Intensity" and at the top by "Greatest Intensity" was obtained during immersion of the subject's non-dominant hand in cold water.
Time Frame: Every 15 seconds during immersion of hand in cold water for up to 5 minutes at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aprepitant | Inert Powder
Number analyzed (Participants) | 16 | 16
units on a scale | 85.8 (16.2) | 81.9 (14.8)

3. Primary Outcome: Unpleasantness of Breathlessness
Description: Time-weighted averages of unpleasantness of breathlessness.
  Subject rating of unpleasantness of breathlessness was obtained at 1 minute intervals during RLB on a 100 mm Visual Analog Scale anchored at the bottom by "No Unpleasantness" and at the top by "Greatest Unpleasantness".
Time Frame: At 1 minute intervals during Resistive Load Breathing at Period 1 (Day 3 or 4) and Period 2 (Day 5, 6 or 7)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Inert Powder: Capsule containing insert powder
Arm/Group | Aprepitant | Inert Powder
Number analyzed (Participants) | 16 | 16
units on a scale | 76.2 (16.7) | 72.2 (20.3)

ADVERSE EVENTS:
Groups:
- Aprepitant: Capsule filled with 125 mg of aprepitant
- Inert Powder: Capsule filled with inert powder
Arm/Group | Aprepitant | Inert Powder
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
1. single dose of aprepitant used
2. clinical diagnosis of chronic bronchitis phenotype of chronic obstructive pulmonary disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No